CLINICAL TRIAL: NCT01544257
Title: Effect of OMT on Length of Stay in a Population of Preterm Infants: RCT Study
Brief Title: Effect of Osteopathic Manipulative Treatment on Length of Stay in Preterms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEO-01
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-02

CONDITIONS: Prematurity
Keywords: Osteopathic manipulative treatment; alternative medicine; complementary medicine; neonatology; neonatal care; prematurity; allied health care
MeSH Terms: conditions — Premature Birth | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMT (Experimental): patients under standard medical care plus OMT.
  Interventions: Other: osteopathic manipulative treatment
- Control (No Intervention): patients under standard medical care plus only osteopathic evaluation
  Interventions: Procedure: Usual care

INTERVENTIONS:
Other: osteopathic manipulative treatment — Patients from this group received osteopathic treatments twice a week for the entire length of stay in the unit.
  Arms: OMT
Procedure: Usual care — Patients from control group received standard care plus osteopathic evaluation only, according to the same schedule as the study group.
  Arms: Control

SUMMARY:
The use of osteopathic manipulative treatment (OMT) in preterm infants has been documented and results from previous studies suggest the association between OMT and length of stay (LOS) reduction, as well as significant improvement in several clinical outcomes. The aim of the present study is to show the effect of OMT on LOS in a sample of premature infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born at age between 29 and 37 weeks
* osteopathic treatment performed < 14 days after birth
* preterms born in the same hospital

Exclusion Criteria:

* gestational age < 29, > 37 weeks;
* osteopathic treatment performed > 14 days after birth;
* newborn transferred to/from other hospital;
* newborn from to HIV seropositive and/or drug addict mother;
* newborn with genetic disorders, congenital abnormalities, cardiovascular abnormalities, neurological disorders, proven or suspected necrotizing enterocolitis with or without gastrointestinal perforation, proven or suspected abdominal obstruction, pre- and/or post-surgery patients, pneumoperitoneum and/or atelectasis.

Ages: 29 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
evaluate the effectiveness of OMT in reducing LOS | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

SECONDARY OUTCOMES:
pre-post difference in weight gain | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, DO, MS, Study Chair — European Institute for Evidence Based Osteopathic Medicine
Locations (1):
- Francesco Cerritelli, Pescara, Italy

REFERENCES:
- [Derived] Cerritelli F, Pizzolorusso G, Ciardelli F, La Mola E, Cozzolino V, Renzetti C, D'Incecco C, Fusilli P, Sabatino G, Barlafante G. Effect of osteopathic manipulative treatment on length of stay in a population of preterm infants: a randomized controlled trial. BMC Pediatr. 2013 Apr 26;13:65. doi: 10.1186/1471-2431-13-65. PMID 23622070